CLINICAL TRIAL: NCT05038787
Title: A Phase 1, Randomized, Investigator- and Participant-Blind, Placebo-Controlled Study of LY3473329 Multiple-Ascending Dosing in Healthy Japanese Participants
Brief Title: A Study of LY3473329 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18097; J2O-JE-EKBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-09-07; First posted 2021-09-09 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3473329 (Experimental): LY3473329 administered orally.
  Interventions: Drug: LY3473329
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3473329 — Administered orally.
  Arms: LY3473329
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3473329 in healthy Japanese participants. The study will also assess how fast LY3473329 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to about 71 days, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined through medical history and physical examination.
* Are males who agree to follow contraception requirements or females not of childbearing potential.
* Are 1st generation Japanese defined as the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.

Exclusion Criteria:

* Have a history or presence of medical illness.
* Have significant history of or current psychiatric disorders.
* Have abnormalities in the 12-lead ECG and blood pressure.
* Have received treatment with siRNA within the past 12 months or any antisense oligonucleotide within the past 6 months for lipoprotein(a) [Lp(a)].

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 43
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3473329 | Predose on Day 1 through Day 43
  PK: AUC of LY3473329
PK: Maximum Concentration (Cmax) of LY3473329 | Predose on Day 1 through Day 43
  PK: Cmax of LY3473329
PK: Time to Maximum Concentration (Tmax) of LY3473329 | Predose on Day 1 through Day 43
  PK: Tmax of LY3473329

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Altasciences Clinical Los Angeles, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No